CLINICAL TRIAL: NCT01394679
Title: A Multicenter Phase 3 Study Comparing the Diagnostic Accuracy of 99mTc EC DG SPECT/CT Versus 18F FDG PET/CT for Diagnosing and Staging Patients Who Have Clinical and Radiological (CT) Evidence Consistent With a Diagnosis of Lung Cancer
Brief Title: A Phase 3 Study of 99mTC-EC-DG SPECT/CT Versus PET/CT in Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cell>Point LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-05-236
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Recurrent Lung Cancer no treatment within 3 months
MeSH Terms: conditions — Lung Neoplasms | interventions — (99m)Tc ethylenedicysteine-deoxyglucose

STUDY DESIGN:
Intervention Model Description: Patients receive Standard PET imaging with FDG then receive SPECT-CT imaging with investigational EC-DG imaging agent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 18-F-FDG Imaging Agent (Active Comparator): 18 F FDG followed by PET/CT imaging
  Interventions: Drug: 18 F FDG followed by PET/CT imaging
- 99m Tc-EC-DG imaging agent (Experimental): 99m Tc-EC-DG injection followed by SPECT/CT imaging (target of 20-30 mCi of Tc)and < 1 mg EC-DG
  Interventions: Drug: (99m Tc) ECDG (Ethylenedicysteine-Deoxyglucose)

INTERVENTIONS:
Drug: (99m Tc) ECDG (Ethylenedicysteine-Deoxyglucose) — One injection of Technetium-99m Ethylenedicysteine-Deoxyglucose to yield a target dose of 25 mCi (range of 20-30 mCi)by IV push and less than 1 mg of EC-DG
  Arms: 99m Tc-EC-DG imaging agent
Drug: 18 F FDG followed by PET/CT imaging — Single injection of 18 F FDG range of 10-20 mCi
  Arms: 18-F-FDG Imaging Agent

SUMMARY:
The purpose of this study is to determine if the images of the primary lesions of lung cancer and any metastatic lesions seen from the investigational SPECT/CT 99mTC-EC-DG scans are the same as the PET/CT 18F-FDG scans.

DETAILED DESCRIPTION:
1. To demonstrate that SPECT/CT (99mTc EC DG) is not inferior to PET/CT (18F FDG PET/CT) for sensitivity or specificity measures when image interpretation of primary and metastatic lesions are compared against a truth standard in patients with a high likelihood of lung cancer.
2. To expand the patient safety experience using 99mTc EC DG.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or female patient at least 18 years old.
2. The subject must agree at the time of enrollment to have the following procedures:

   * A tissue diagnosis of the primary lesion either prior to enrollment or within 15 days of the PET/CT study but before initiation of therapy
   * A SPECT/CT procedure
   * A baseline DCCT scan
   * A whole-body bone scan
   * A follow-up focused DCCT scan (if indicated)
3. The patient has had a non incisional biopsy demonstrating definitive evidence for lung cancer OR have clinical evidence and CT scan results consistent with a diagnosis of lung cancer. Cytology results confirming lung cancer from a bronchoscope procedure will also be acceptable. A copy of the actual report (biopsy/cytology or CT scan) must be requested by the patient through a medical release form if not already done. The copy must be available to the study doctor within 15 days of the PET imaging study.
4. The patient will not be receiving treatment for lung cancer (surgery, radiation, and/or chemotherapy), or, if the patient has had lung cancer in the past, all previous therapy was completed at least 3 months prior to being enrolled in the study.
5. If a tissue diagnosis of the primary lesion was not done prior to enrollment, the patient must agree to have a tissue diagnosis of the primary lesion within 15 days of the PET/CT study but prior to initiation of therapy, independent of the PET/CT results.
6. The patient must be referred for a PET/CT scan on the basis of clinical and radiological (CT) evidence for a diagnosis of lung cancer.
7. The patient will have an Eastern Co-operative Oncology Group (ECOG) performance rating < or = 2.
8. The patients will be males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy).
9. Females of childbearing potential and males with female sexual partners of childbearing potential must agree to use one of the following acceptable birth control methods:

   1. Surgically sterile (hysterectomy or bilateral oophorectomy)
   2. Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation - documentation is required)
   3. Intrauterine device (IUD) in place for at least 3 months
   4. Double-barrier method (condom and diaphragm) with spermicide for at least 14 days prior to screening and through study completion
   5. Stable hormonal contraceptive (oral, topical, vaginal or implanted/injected) for at least 3 months prior to study and through study completion
   6. Abstinence
   7. Single-barrier method for at least 14 days prior to screening and through study completion for vasectomized males or females with vasectomized partners
10. The patient will have fasting blood glucose of < 200 mg/dL at screening.
11. The patient will have reported clinical symptoms consistent with a diagnosis of lung cancer.
12. The patient must be able to tolerate SPECT/CT and PET/CT imaging. This includes:

    1. lying in the same position without moving for approximately 45 minutes
    2. able to tolerate a confined area (ie, not claustrophobic)
    3. ability to hold their arms overhead for approximately 45 minutes
13. The patient must be able to fast and/or follow diet restrictions prior to SPECT/CT and PET/CT imaging.
14. Patients must fast for at least 6 hours prior to the injection for the study.
15. The patient must be able to eat a high protein/low carbohydrate meal as the last meal before SPECT/CT and PET/CT imaging. However, if the site has its own standard of care requirements for fasting and/or diet restrictions for PET as an alternative to this recommendation, the same fasting and/or diet restrictions used for PET imaging should be applied for the SPECT imaging.
16. The patient must be able to make the scheduled appointments within the designated time windows (PET/CT imaging within 7 days of qualifying for the study, the second imaging session with SPECT/CT imaging 1-15 days after the initial imaging visit, with at least 24 hours between PET/CT and SPECT/CT imaging).
17. The patient must have safety laboratory values that, in the opinion of the Investigator, do not place the patient at undue risk if the patient were to participate in the study. This includes (but is not limited to):

    1. alanine aminotransferase < or = 2.5 × ULN
    2. aspartate aminotransferase < or = 2.5 × ULN
    3. creatinine < or = 2.5 × ULN
    4. bilirubin < or = 2.0 × ULN
18. The patient must be able to understand and provide signed informed consent.
19. Females of childbearing potential must have a negative urine or serum β-hCG pregnancy test at screening.

Exclusion Criteria:

1. Any clinically significant safety concerns (laboratory, EKG, physical examination, other) that, in the opinion of the Investigator, would place the patient at undue risk if the patient were to participate in the study.
2. The patient is undergoing any current treatment for cancer (radiation therapy, surgery, or chemotherapy).
3. The patient is diabetic with insulin dependence. (Patients who have known insulin dependence for diabetes can be included in the study if the standard of care protocol in place at the clinical site provides for the management of the patient's glucose level sufficiently to allow the PET/CT imaging to be performed. The same glucose management used for the PET/CT imaging should be applied to the SPECT/CT imaging procedures. A waiver will be required to be completed by the clinical site and approved by the sponsor or designee.)
4. The patient's weight is above the SPECT/CT and PET/CT table weight limit.
5. The patient has a known hypersensitivity to EC DG or FDG or similar compounds including any of the inactive ingredients.
6. The patient has a known or suspected pregnancy, lactation or planned pregnancy (females and male partners).
7. The patient has clinically significant mental illness (to be determined by the Investigator).
8. The patient has exposure to any investigational agent within 30 days prior to the screening visit or is participating in an ongoing clinical study. (This criterion can be overruled by the Principal Investigator with appropriate documentation of the reason for the exception.)
9. The patient has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy:Comparison of 99mTc-EcC-DG SPECT/CT images to 18F-FDG PET/CT images of primary lung cancer lesion and metastatic lesions | Images will be compared at the core image lab at approximately every 4 to 6 weeks
  To demonstrate that SPECT/CT (99mTc EC DG) is not inferior to PET/CT (18F FDG PET/CT) for sensitivity or specificity measures when image interpretation of primary and metastatic lesions are compared against a truth standard in patients with a high likelihood of lung cancer.

SECONDARY OUTCOMES:
Safety:Through Adverse Event Collection | From 99m-Tc-EC-DG injection up to 90 days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Phurrough, BS, Study Director — Consultanat
Locations (1):
- Decatur Memorial Hospital, Decatur, Illinois, United States